CLINICAL TRIAL: NCT05061901
Title: Randomized Crossover 2 Period Single Dose Bioequivalence Study of 2 Formulations Lisinopril Tab. 20mg (Pharmtechnology LLC,Belarus) and Zestril® Tab. 20mg (Avara Reims Pharmaceutical Services, France) in Healthy Volunteers Under Fasting Conditions
Brief Title: Bioequivalence Study of Two Formulations of Lisinopril Tablet 20 mg in Healthy Volunteers Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmtechnology LLC (Industry)
Collaborators: ClinPharmInvest, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: LZNP-2020-CPI-FRMT
Record Dates: First submitted 2021-09-20; First posted 2021-09-30 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Bioequivalence
MeSH Terms: interventions — Lisinopril

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence TR (Other): 19 subjects assigned to the sequence TR will receive a single 20 mg dose of the test product Lisinopril (1 x 20 mg tablet), marked as T in the sequence, in Period 1 and a single 20 mg dose of the reference product Zestril® (1 x 20 mg tablet), marked as R in the sequence, in period 2. These treatments will be administered orally with approximately 200 mL of water, in the morning, following a 10-hour overnight fast. The tablet must be swallowed whole and must not be chewed or broken.
  Interventions: Drug: Lisinopril tablet 20 mg
- Sequence RT (Other): 19 subjects assigned to the sequence RT will receive a single 20 mg dose of the reference product Zestril® (1 x 20 mg tablet), marked as R in the sequence, in Period 1 and a single 20 mg dose of the test product Lisinopril (1 x 20 mg tablet), marked as T in the sequence, in period 2. These treatments will be administered orally with approximately 200 mL of water, in the morning, following a 10-hour overnight fast. The tablet must be swallowed whole and must not be chewed or broken.
  Interventions: Drug: Zestril® tablet 20 mg

INTERVENTIONS:
Drug: Lisinopril tablet 20 mg — Lisinopril is manufactured by Pharmtechnology LLC, Belarus. Each tablet contains 20 mg of lisinopril.
  Other Names: The test product
  Arms: Sequence TR
Drug: Zestril® tablet 20 mg — Zestril® is manufactured by Avara Reims Pharmaceutical Services, France. Each tablet contains 20 mg of lisinopril.
  Other Names: The reference product
  Arms: Sequence RT

SUMMARY:
This is an open-labeled (laboratory blinded), randomized, two period, single-center, crossover, comparative study, where each participant will be randomly assigned to the reference (Zestril®, 20 mg) or the test (Lisinopril, 20 mg) formulation in each period of study (sequences Test-Reference (TR) or Reference-Test (RT)), in order to evaluate if both formulations are bioequivalent

ELIGIBILITY:
Inclusion Criteria:

1. Healthy caucasian men and women aged between 18 to 45 years
2. Verified diagnosis "healthy" according to the anamnesis data and the results of standard clinical, laboratory and instrumental examination methods, physical examination and anamnestic examination
3. The results of an X-ray or fluorographic examination of the chest organs within the normal range (the results of an examination carried out within 12 months before the start of the study may be provided)
4. Satisfactory tolerance of the orthostatic test (the range of increase in heart rate when moving from a prone position to a standing position within 12 - 18 beats per minute)
5. Body mass index 18.5-30 kg/m² according to Quetelet's weight-height index
6. For female subject:

   * the results of the examination of the mammary glands (palpation or mammography) within the normal range according to the data obtained within 12 months before the start of the study;
   * non-breastfeeding women;
   * negative pregnancy test;
   * adherence to reliable methods of contraception for female of childbearing potential: sexual continence, or condom + spermicide, or diaphragm + spermicide, started at least 14 days before the first dose of the study drug; intrauterine contraception is also a reliable method of contraception, installed at least 4 weeks before taking the study drugs in the first period;
   * сonsent to use these methods of contraception within 30 days after taking the drug in the second period;
   * women who do not use acceptable methods of contraception, if they are considered incapable of childbearing, will also be able to participate in the study: women who have undergone a hysterectomy or tubal ligation, women with a clinical diagnosis of infertility, and women who are in menopause (at least a year without menstruation in the absence of alternative pathologies that may cause the cessation of menstruation);
   * in case of using contraceptives (injectable and oral hormonal contraceptives, subcutaneous hormonal implants or intrauterine hormonal therapeutic systems), the latter should be canceled at least 60 days before taking the drug in the first period;

Exclusion Criteria:

1. burdened allergic history, hypersensitivity to any ACE inhibitors, including lisinopril or excipients that are part of any of the investigational drugs, or intolerance to these components;
2. a history of angioedema, including associated with the use of ACE inhibitors, idiopathic angioedema, hereditary angioedema;
3. clinically significant pathologies of the cardiovascular, bronchopulmonary, neuroendocrine systems, as well as diseases of the gastrointestinal tract, liver, kidneys and blood;
4. other diseases that, in the opinion of the researcher, may affect the absorption, distribution, metabolism or excretion of both drugs, or increase the risk of negative consequences for the volunteer;
5. the presence of mental disorders, including a history;
6. surgical interventions on the gastrointestinal tract, with the exception of appendectomy;
7. acute infectious diseases that ended less than 4 weeks before taking the drug in the first period;
8. dehydration due to diarrhea, vomiting or other reason within the last 24 hours before taking the drug in the first period of the study;
9. clinically significant abnormalities on the ECG, the level of systolic blood pressure (SBP) measured in the sitting position at the time of screening ≤ 100 mm Hg or ≥ 130 mm Hg and / or diastolic blood pressure (DBP) ≤ 60 mm Hg or ≥ 85 mm Hg;
10. heart rate less than 60 beats/min or more than 90 beats/min at the time of screening, respiratory rate less than 12 or more than 18 per minute at the time of screening, body temperature below 36.0 ° C or above 37.0 °C at the time of screening;
11. unsatisfactory tolerance of the orthostatic test (the difference between the heart rate values when moving from a prone position to a standing position is less than 12 or more than 18 beats per minute;
12. the use of injectable and oral hormonal contraceptives, subcutaneous hormonal implants or intrauterine hormonal therapeutic systems and other hormonal contraceptives for 60 days before taking the drug in the first period;
13. use of any drugs including herbs and food additives, vitamins that can have a significant effect on the PK of lisinopril or data on the effect of which on the pharmacokinetics of lisinopril are unknown, as well as question the characterization of the volunteer as healthy, less than 14 days before taking the drug in the first period;
14. donation of plasma or blood (450 ml or more) less than 2 months before taking the drug in the first period;
15. consumption of caffeine and xanthine-containing drinks and products (tea, coffee, chocolate, cola, etc.), products containing poppy seeds, less than 48 hours before taking the drug in the first period;
16. consumption of alcohol and alcohol-containing foods and beverages less than 48 hours before taking the drug in the first period;
17. use of citrus fruits (including grapefruit and grapefruit juice) and cranberries (including juices, fruit drinks, etc.) less than 7 days before taking the drug in the first period;
18. intake of more than 10 units alcohol per week (1 unit of alcohol is equivalent to 500 ml of beer, 200 ml of dry wine or 50 ml of spirits ethyl 40%) or history of alcoholism, drug addiction, drug abuse;
19. inability to refrain from intensive physical activity and contact sports less than 24 hours before taking the drug in the first period;
20. smoking more than 10 cigarettes per day less than 24 hours before taking the drug in the first period;
21. participation in other clinical trials of drugs less than 3 months before taking the drug in the first period;
22. test positive for syphilis, hepatitis B, hepatitis C or HIV at the time of screening;
23. positive pregnancy test at screening;
24. breastfeeding;
25. positive test for alcohol in exhaled air at screening;
26. positive urinalysis for the content of narcotic and potent substances during screening (opiates, morphine, barbiturates, benzodiazepines, cannabinoids/marijuana);
27. the value of standard laboratory and instrumental parameters that go beyond the reference values;
28. lack of intention of volunteers to comply with the Protocol requirements throughout the course of the study and/or lack, in the opinion of the Investigator, of the volunteers' ability to understand and evaluate the information on this study as part of the informed consent form signing process, in particular regarding the expected risks and possible discomfort;
29. tattooing and piercing within 30 days prior to first drug administration;
30. difficulty swallowing tablets;
31. difficulty with taking blood;

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2021-11-06 (Actual); Study Completion 2021-11-06 (Actual)

PRIMARY OUTCOMES:
Cmax of lisinopril in plasma after administration of the test and the reference products. | Time points 0.00 (prior to each drug administration) and 1.00, 2.00, 3.00, 4.00, 5.00, 6.00, 6.50, 7.00, 7.50, 8.00, 9.00, 10.00, 12.00, 16.00, 20.00, 24.00, 36.00, 48.00, 72.00 hours after each drug administration.
  Maximum observed concentration in plasma.
AUC0-t of lisinopril in plasma after administration of the test and the reference. | Time points 0.00 (prior to each drug administration) and 1.00, 2.00, 3.00, 4.00, 5.00, 6.00, 6.50, 7.00, 7.50, 8.00, 9.00, 10.00, 12.00, 16.00, 20.00, 24.00, 36.00, 48.00, 72.00 hours after each drug administration.
  Cumulative area under the concentration time curve calculated from 0 to time of last observed quantifiable concentration (TLQC) using the linear trapezoidal method.

SECONDARY OUTCOMES:
Tmax of lisinopril in plasma after administration of the test and the reference products. | Time points 0.00 (prior to each drug administration) and 1.00, 2.00, 3.00, 4.00, 5.00, 6.00, 6.50, 7.00, 7.50, 8.00, 9.00, 10.00, 12.00, 16.00, 20.00, 24.00, 36.00, 48.00, 72.00 hours after each drug administration.
  Tmax of lisinopril in plasma after administration of the test and the reference products.
TLQC of lisinopril in plasma after administration of the test and the reference products. | Time points 0.00 (prior to each drug administration) and 1.00, 2.00, 3.00, 4.00, 5.00, 6.00, 6.50, 7.00, 7.50, 8.00, 9.00, 10.00, 12.00, 16.00, 20.00, 24.00, 36.00, 48.00, 72.00 hours after each drug administration.
  Time of last observed quantifiable concentration.
AUC0-INF of lisinopril in plasma after administration of the test and the reference products. | Time points 0.00 (prior to each drug administration) and 1.00, 2.00, 3.00, 4.00, 5.00, 6.00, 6.50, 7.00, 7.50, 8.00, 9.00, 10.00, 12.00, 16.00, 20.00, 24.00, 36.00, 48.00, 72.00 hours after each drug administration.
  Area under the concentration time curve extrapolated to infinity, calculated as AUC0-t + ĈLQC (the predicted concentration at time TLQC) / λZ (apparent elimination rate constant).
Residual area of lisinopril in plasma after administration of the test and the reference products. | Time points 0.00 (prior to each drug administration) and 1.00, 2.00, 3.00, 4.00, 5.00, 6.00, 6.50, 7.00, 7.50, 8.00, 9.00, 10.00, 12.00, 16.00, 20.00, 24.00, 36.00, 48.00, 72.00 hours after each drug administration.
  Extrapolated area (i.e. percentage of AUC0-INF due to extrapolation from TLQC to infinity).
Time point where the log-linear elimination phase begins (TLIN) of lisinopril in plasma after administration of the test and the reference products. | Time points 0.00 (prior to each drug administration) and 1.00, 2.00, 3.00, 4.00, 5.00, 6.00, 6.50, 7.00, 7.50, 8.00, 9.00, 10.00, 12.00, 16.00, 20.00, 24.00, 36.00, 48.00, 72.00 hours after each drug administration.
  Time point where the log-linear elimination phase begins.
λZ of lisinopril in plasma after administration of the test and the reference products. | Time points 0.00 (prior to each drug administration) and 1.00, 2.00, 3.00, 4.00, 5.00, 6.00, 6.50, 7.00, 7.50, 8.00, 9.00, 10.00, 12.00, 16.00, 20.00, 24.00, 36.00, 48.00, 72.00 hours after each drug administration.
  Apparent elimination rate constant, estimated by linear regression of the terminal linear portion of the log concentration versus time curve.
Terminal elimination half-life (Thalf) of lisinopril in plasma after administration of the test and the reference products. | Time points 0.00 (prior to each drug administration) and 1.00, 2.00, 3.00, 4.00, 5.00, 6.00, 6.50, 7.00, 7.50, 8.00, 9.00, 10.00, 12.00, 16.00, 20.00, 24.00, 36.00, 48.00, 72.00 hours after each drug administration.
  Terminal elimination half-life, calculated as ln(2)/λZ.
Number of treatment-emergent adverse events for the test and the reference products. | Time points 0.00 (prior to each drug administration) and 1.00, 2.00, 3.00, 4.00, 5.00, 6.00, 6.50, 7.00, 7.50, 8.00, 9.00, 10.00, 12.00, 16.00, 20.00, 24.00, 36.00, 48.00, 72.00 hours after each drug administration.
  The safety population will include all subjects who received at least one dose of the test or the reference product. Any significant changes will be recorded as treatment-emergent adverse events only if they are judged clinically significant by the qualified investigator or delegate.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Khokhlov, Principal Investigator — ClinPharmInvest, LLC
Locations (1):
- Private healthcare institution "Clinical Hospital "RZD-Medicine" of the city of Yaroslavl", Yaroslavl, Yaroslavl Oblast, Russia